CLINICAL TRIAL: NCT00970359
Title: Reacquisition of RAI Uptake of RAI-Refractory Metastatic Thyroid Cancers by Pretreatment With the Selective MEK Inhibitor AZD6244: A Pilot Study
Brief Title: Reacquisition of Radioactive Iodine (RAI) Uptake of RAI-Refractory Metastatic Thyroid Cancers by Pretreatment With the Selective MEK Inhibitor AZD6244
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-048
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Thyroid Cancer
Keywords: thyroid; metastases; AZD6244; 09-048
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases; Neoplasm Metastasis | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pts with thyroid cancer with and without BRAF mutation (Experimental): Patients receive selumetinib orally (PO) twice daily (BID) for 4 weeks. Within 1 month, patients with adequate RAI uptake may receive 131I per standard of care and continue selumetinib until 2 days following 131I.
  Interventions: Biological: AZD6244

INTERVENTIONS:
Biological: AZD6244 — Within 1 week of starting the study: Low iodine diet
  The patient will receive three bottles of capsules containing the drug AZD6244. Each capsule contains 25 milligrams of AZD6244. They will take 3 capsules orally, by mouth twice a day for 4 weeks. AZD6244 should be taken on an empty stomach (either one hour before or 2 hours after meals). AZD6244 capsules should be taken with water only. Lesional dosimetry with iodine-124 PET will be done twice, at the beginning and at the end of the study. This is done the same way that a radioactive iodine scan is done and is spread out over 5 days. It requires injection with human recombinant TSH (Thyrogen) on day 1 and 2, as well as blood tests on day 1 and day 5. On day 3, you will receive the iodine-124 in form of an oral drink, and the PET scan will be obtained on day 5. You will need to follow a low iodine diet starting 5 days before and throughout the process.

SUMMARY:
The purpose of this study is to find out if the drug AZD6244 can improve the radioactive iodine uptake by the patient's metastatic thyroid cancer. The investigator will also be testing the tumor specimen taken at the time of your surgery for specific genetic changes to see if one of them in particular (the BRAF oncogene) makes your cancer more likely to become sensitive to radioactive iodine after treatment with the drug.

The investigators want to find out if AZD6244 helps to increase the entry of radioactive iodine into thyroid cancer cells that have spread and are resistant to radioactive iodine therapy, especially if they have the BRAF mutation. To measure how much iodine can enter your cancer, the investigators will use iodine-124, a different form of radioactive iodine. Iodine-124 allows the investigators to measure precisely how much radioactivity can enter the cancer cells, whereas iodine-131 does not. The process of scanning with iodine-124 is called "lesional dosimetry". Iodine-124 is an investigational agent approved by the FDA (Food and Drug Administration) for use in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = to 18 years-old
* Patients must have histopathologically confirmed at MSKCC differentiated thyroid carcinoma of follicular cell origin (D-TC-FCO), which includes papillary, follicular, or Hürthle cell histology, along with their respective variants.
* Pathology specimen from the original tumor (thyroid) and/or metastases must be available for genotyping.
* RAI-refractory metastatic disease on structural imaging, defined as any one of the following (as described in MSKCC protocol 08-066):

  * index metastatic lesion non-RAI avid on a diagnostic RAI scan performed up to 2 years prior to enrolment in the current study, OR
  * RAI-avid metastatic lesion which remained stable in size or progressed despite RAI treatment 6 months or more prior to entry in the study. Lesions will be assessed by 2 independent observers in nuclear medicine and in endocrinology. There is no minimal size limit for the index lesion.
* Patients with FDG avid lesions
* Evaluable disease by RECIST
* Preliminary reproductive toxicology data indicate that AZD6244 can have adverse effects on embryofetal development and survival at dose levels that do not induce maternal toxicity in mice. For this reason, female patients will need to be post-menopausal or with negative serum pregnancy test if pre-menopausal. Patients of childbearing potential must agree to employ adequate contraception throughout the study.
* ANC > 1500 per mm3, platelets > 100,000 per mm3, and hemoglobin > 9 g/dL
* ALT/SGOT and AST/SGPT ≤ 2.5 X upper limit of normal (ULN)
* Bilirubin ≤ 1.5 X ULN
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patient with chronic renal insufficiency, as defined initially by an estimated creatinine clearance of < 30 ml/minute calculated using the Cockcroft and Gault equation: (140 - age in years) X (weight in kg) X (0.85 if female)/72 X serum Cr. If estimated creatinine clearance is < 30 ml/min, a 24 hour urine creatinine clearance may be collected and a patient would be eligible if the creatinine clearance is >30 ml/min.
* Patients unable to follow a low iodine diet, patients requiring medication with high content in iodide (amiodarone), or patients receiving IV iodine containing contrast as part of radiographic procedure.
* Patients with clinically significant cardiovascular disease as defined by the following:

  * LVEF < institutional LLN
  * New York Heart Association grade III or greater congestive heart failure
  * uncontrolled hypertension, defined as systolic blood pressure > 180 mmHg OR diastolic blood pressure > 105 mmHg, on at least 2 repeated determinations on separate days within past 3 months
  * Uncontrolled coronary artery disease, angina, congestive heart failure, or ventricular arrhythmia requiring acute medical management.
* Patient with known hypersensitivity to Thyrogen (human recombinant thyrotropin).
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women will be ineligible; breast feeding should be discontinued if the mother is treated with AZD6244.
* Brain metastases or spinal cord compression unless treated and stable (for at least 3 months) off steroids.
* Mean QTc interval >450 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ho, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Ho AL, Grewal RK, Leboeuf R, Sherman EJ, Pfister DG, Deandreis D, Pentlow KS, Zanzonico PB, Haque S, Gavane S, Ghossein RA, Ricarte-Filho JC, Dominguez JM, Shen R, Tuttle RM, Larson SM, Fagin JA. Selumetinib-enhanced radioiodine uptake in advanced thyroid cancer. N Engl J Med. 2013 Feb 14;368(7):623-32. doi: 10.1056/NEJMoa1209288. PMID 23406027
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZD6244
Started | 24
Completed | 20
Not Completed | 4
Not completed — Not Treated | 4

BASELINE CHARACTERISTICS:
Arm/Group | AZD6244
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Whose Tumor(s) Acquire an Increased Propensity for Iodine Uptake as Detected on Iodine-124 Positron Emission Tomography Scan
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | AZD6244
Number analyzed (Participants) | 20
participants
  New and/or increase | 12
  Remained the same or less | 8

2. Primary Outcome: Tumor Response Defined as Either a Complete Response or Partial Response
Description: as defined by the RECIST v1.1 criteria Descriptive statistics will be used to summarize the data.
Time Frame: 6 months
Population: Only patients treated with radioiodine.
Measure: Number; unit: participants
Arm/Group | AZD6244
Number analyzed (Participants) | 8
participants
  Partial Response | 5
  Stable Disease | 3

3. Secondary Outcome: Change From Baseline in Serum Thyroglobulin Levels After Treatment With 131I
Description: Will perform a Wilcoxon signed rank test for paired samples to compare the serum thyroglobulin level before and after 131I treatment in the subset of patients treated with 131I following AZD6244.
Time Frame: At 2 months and 6 months after Radioiodine administration
Population: Only patients treated with Radioiodine.
Measure: Mean (Full Range); unit: percentage of reduction of levels
Arm/Group | AZD6244
Number analyzed (Participants) | 8
percentage of reduction of levels
  at 2 months | 89 [74.4 to 99.9]
  at 6 months | 80 [5.1 to 100]

ADVERSE EVENTS:
Arm/Group | AZD6244
Serious Adverse Events (participants affected / at risk) | 2/24
Other Adverse Events (participants affected / at risk) | 11/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6244 (N=24)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6244 (N=24)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes